CLINICAL TRIAL: NCT02412917
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Comparative Study of FV-100 vs. Valacyclovir for the Prevention of Post-Herpetic Neuralgia and Treatment of Acute Herpes Zoster Associated Pain
Brief Title: A Comparative Study of FV-100 vs. Valacyclovir for the Prevention of Post-Herpetic Neuralgia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: ContraVir Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: ContraVir (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CTRV-FV-2-007
Record Dates: First submitted 2015-03-23; First posted 2015-04-09 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Shingles; Herpes Zoster; Postherpetic Neuralgia
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic | interventions — FV-100; Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FV-100 400 mg QD (Experimental): FV-100 400mg QD
  Interventions: Drug: FV-100
- FV-100 400mg BID (Experimental): FV-100 400mg BID(total daily dose of 800mg)
  Interventions: Drug: FV-100
- valacyclovir (Active Comparator): valacyclovir 1000mg TID
  Interventions: Drug: valacyclovir

INTERVENTIONS:
Drug: FV-100 — antiviral nucleoside analog
  Other Names: antiviral nucleoside analog
  Arms: FV-100 400 mg QD; FV-100 400mg BID
Drug: valacyclovir — antiviral nucleoside analog
  Other Names: valtrex
  Arms: valacyclovir

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-group, active controlled comparative study of the safety and efficacy of 2 dosing regimens of FV-100 versus valacyclovir administered for 7 days in subjects with uncomplicated AHZ(acute herpes zoster).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group, active controlled comparative study of the safety and efficacy of 2 dosing regimens of FV-100 versus valacyclovir administered for 7 days in subjects with uncomplicated AHZ(acute herpes zoster). Subjects diagnosed with uncomplicated AHZ within 72 hours of lesion appearance and worst pain of 4 or greater at day 1, will be randomized (1:1:1) to one of three treatment groups and will begin study treatment at the Day 1 visit(within 72 hours of AHZ lesion appearance) to either: 1. FV-100 400mg QD, 2. FV-100 400mg BID(total daily dose of 800mg), or 3. Valacyclovir 1000mg 3 times a day for a total daily dose of 3000mg. Subjects will be monitored for adverse events through day 21. Efficacy assessments for lesion status and AHZ pain are captured til day 120.

ELIGIBILITY:
Inclusion Criteria:

* Receive a clinical diagnosis of uncomplicated AHZ as evidenced by a unilateral dermatomal rash
* Have zoster-related pain
* Are able to be randomized and receive their first dose within approximately 120 hours from appearance of rash

Exclusion Criteria:

* Have multidermal or disseminated AHZ
* Have facial, ophthalmologic or oral manifestations
* Have received Zostavax

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2015-06; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The incidence of post-herpetic neuralgia(PHN) following treatment with 2 dose regimens of FV-100 compared to valacyclovir. | Day 1 to Day 120
  efficacy measure

SECONDARY OUTCOMES:
Acute herpes zoster associated pain, as measured by Zoster Brief Pain Inventory(ZBPI) | Day 1 to Day 120
  efficacy measure
The effect on lesion formation and healing of 2 dose regimens of FV-100 compared to valacyclovir | Day 1 to Day 120
  efficacy measure
The number and classification of adverse events in 2 dosing regimens of FV-100 | Day 1 to Day 120
  Safety measure
The pharmacokinetic profile of the active metabolite of FV-100 after 7 days of dosing at 400mg QD versus compared with 400mg BID | Day 1 to Day 120
  Pharmacokinetic

CONTACTS AND LOCATIONS:
Overall Officials: John Sullivan-Bolyai, Study Director — CMO
Locations (1):
- TX, Webster, Texas, United States